CLINICAL TRIAL: NCT00292773
Title: The Effect of Weight Reduction Surgery on Ovarian Function in Obese Anovulatory Patients
Brief Title: Weight Reduction Surgery and Ovarian Function
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Prof Simon Heller, Sheffield Teaching Hospitals NHS Foundation Trust
Other Study IDs: STH14006
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Anovulation; Obesity
Keywords: Anovulation; Obesity; bariatric surgery
MeSH Terms: conditions — Anovulation; Obesity

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: weight reduction minimal access surgery — Patients will be offered laparoscopic gastric bypass surgery by Mr Roger Ackroyd, in line with the current recommendation for gastric surgery according to NICE guidelines i.e. patients with a BMI over 40 or a BMI over 35 with at least one co-morbidity. Patients will be reviewed monthly for six months.

SUMMARY:
This study will investigate the role of weight reduction surgery on the reproductive performance of obese women with ovulation problems. It is hypothesized that surgery offered when other methods of weight reduction have failed, may help restore ovulation.

DETAILED DESCRIPTION:
We aim to recruit 30 patients suffering from chronic anovulation, with a body mass index of 35 or more, who failed to achieve weight reduction with other methods such as orlistat, metformin, diet and exercise.

Patients will be approached by one of the investigators in the infertility clinics and the assisted conception unit of the Royal Hallamshire hospital. Consent will be obtained by one of the designated investigators. The consent form has been designed in accordance with the guidelines of the central office for research and ethics committees (COREC). A patient information leaflet will be supplied and has been designed according to the COREC guidelines.

Patients will have a baseline history, clinical examination, hormonal profile (FSH/LH, fasting Insulin/glucose ratio, androgen profile, day 21 serum progesterone, serum leptin and ghrelin levels) ultrasound examination (ovarian volume and antral follicle count), including Doppler blood flow study (ovarian stromal velocity).

Patients will be offered laparoscopic gastric bypass surgery by Mr Roger Ackroyd, in line with the current recommendation for gastric surgery according to NICE guidelines i.e. patients with a BMI over 40 or a BMI over 35 with at least one co-morbidity. Patients will be reviewed monthly for six months. At each visit the following will be recorded:

1. Weight, menstrual diary.
2. Hormonal profile (FSH/LH, fasting Insulin/glucose ratio, androgen profile, day 21 serum progesterone, serum leptin and ghrelin levels).
3. Doppler of ovarian stroma (Pulsitility index, Peak velocity), ovarian volume and antral follicle count
4. Review of symptomatology especially androgenic symptoms.

End point:

Completion of six months follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Anovulation or irregular ovulation as determined by the following clinical or laboratory features:

   * Clinical:

     i. Irregular cycles (not 25-35 days) ii. Amenorrhoea (more than six months).
   * Biochemical: Day 21 or midleuteal serum progesterone of less than 30mmol/l.
2. BMI of 35 or more.
3. Age between 18 and 45.

Exclusion Criteria:

1. Contraindication for bypass surgery:

   i. Medically unfit ii. Psychologically unfit iii. Strong family history of gastric cancer
2. Insulin dependant diabetes or patients on oral hypoglycaemics. Insulin resistance and impaired glucose tolerance however, are not exclusion criteria.
3. Concomitant endocrine disorders including thyroid disease and Cushing syndrome.
4. Patients on steroid therapy.
5. Patients who have had one or both ovaries removed.
6. Biochemical evidence of ovarian failure i.e. FSH of 20 IU or more.
7. Patients who have had hysterectomy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese anovulatory women.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor TC Li, FRCOG,MD, Study Chair — STH; Professor William Ledger, FRCOG,D Phil, Study Chair — Sheffield University
Locations (1):
- Jessop Wing, Royal Hallamshire Hospital, Sheffield, United Kingdom